CLINICAL TRIAL: NCT01197625
Title: Trial of Vaccine Therapy in Curative Resected Prostate Cancer Patients Using Autologous Dendritic Cells Loaded With mRNA From Primary Prostate Cancer Tissue, hTERT and Survivin
Brief Title: Vaccine Therapy in Curative Resected Prostate Cancer Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Knut Halvor Bjøro Smeland, MD PhD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC-005
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer
Keywords: Vaccination treatment, dendritic cells
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DC-vaccine (Experimental)
  Interventions: Biological: Dendritic cell vaccine

INTERVENTIONS:
Biological: Dendritic cell vaccine — Autologous Dendritic Cells Loaded With mRNA From Primary Prostate Cancer Tissue, hTERT and Survivin

SUMMARY:
In this study the investigators will include patients with high risk of PSA relapse scheduled to receive curative surgical treatment. This include patients with high Gleason score (9-10) or micrometastatic disease (tumor cells detected in specimens obtained from bone marrow). They are scheduled for regular follow-ups with PSA measurements. We have previously published that some patients with metastatic prostate cancer may respond to DC-vaccination with tumor mRNA, with a decrease in PSA. PSA response is related to immunological response. Patients receiving DC-vaccination may have a reduced risk of PSA relapse or increased time to PSA relapse. Previous experience with different DC-vaccine protocols in our hospital has resulted in only minor side-effects (grade 1-2 fever, rubor, fatigue, local swelling or pain).

ELIGIBILITY:
Inclusion Criteria:

* Radical prostatectomy. Preferably accessible tumor tissue with enough volume and quality for vaccine production (extraction of tumor mRNA).
* Pathological stage pT2 - pT3b and Gleason score 7B-10, pN0, pN+ or pNx.
* Must be ambulatory with an ECOG performance status 0 or 1.
* Tumor cells detected in bone-marrow samples (micrometastatic disease). Patients with Gleason score 9-10 or pT3b Gleason score 8 may also be included with negative bone-marrow aspiration. Bone-marrow aspirates and plasma for microRNA will be obtained before start of surgery.
* Must be at least 18 years of age and less than 75 years.
* PSA < 0.2 µg/L within 6 weeks after surgery.
* Must have lab values as the following:

ANC ≥ 1.5 x 109/L; Platelets ≥ 100 x 109/L; Hb ≥ 9 g/dL (≥ 5.6 mmol/L); Creatinine ≤ 140 μmol/L (1.6 mg/dL)- if borderline, the creatinine clearance ≥ 40 mL/min; Bilirubin within the upper limit of normal; ASAT and ALAT ≤ 2.5 the upper limit of normal; Albumin levels above lower normal value

* No metastasis on bone scans or MRI, last 3 months before inclusion.
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Previous treatment with LHRH (Luteinizing Hormone-Releasing Hormone) agonist.
* Previous anti-androgen treatment (Casodex).
* History of prior malignancy within the last 5 years, with the exception of curatively treated basal cell carcinoma.
* Active infection requiring antibiotic therapy.
* Significant cardiac or other medical illness that would limit activity or survival, such as severe congestive heart failure, unstable angina, or serious cardiac arrhythmia.
* Adverse reactions to vaccines such as asthma, anaphylaxis or other serious reactions.
* History of immunodeficiency or autoimmune disease such as rheumatoid arthritis, systemic lupus erythematosus, scleroderma, polymyositis-dermatomyositis, juvenile onset insulin dependent diabetes, or a vasculitic syndrome.
* Positive testing for syphilis (treponema pallidum), HIV, Hepatitis B and C
* Use of systemic glucocorticoids.
* Any reason why, in the opinion of the investigator, the patient should not participate.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-09; Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure defined by two different measurement of PSA levels >0.5 µg/L with minimum of 4 weeks interval in patients receiving treatment | From date of vaccination until the date of first documented treatment failure, assessed up to 8 years

SECONDARY OUTCOMES:
Safety and toxicity of vaccination. Evaluation of immunological response. | Up to 8 years after vaccination

OTHER OUTCOMES:
Efficacy Outcome Measure Efficacy Outcome Measure Percentage of patients with a second positive bone marrow examination at the End of Treatment | Up to 36 month
Time to PSA levels > 0.5 μg/L defined by two different measurement of PSA levels > 0.5 μg/L with minimum of 4 weeks interval in patients included by signing the informed concent form, but not receiving treatment | From date of vaccination until the date of first documented treatment failure, assessed up to 8 years
  Pathological stage pT2 - pT3b and Gleason score 7B-8, pN0, pN+ or pNx. Negative bone marrow examination

CONTACTS AND LOCATIONS:
Overall Officials: Knut HB Smeland, M.D PhD, Principal Investigator — Oslo University Hospital - Norwegian Radium Hospital
Locations (1):
- The Norwegian Radium Hospital, Department of Clinical Cancer Research, Oslo, Norway

REFERENCES:
- See also: Hospital's website — https://oslo-universitetssykehus.no